CLINICAL TRIAL: NCT07199504
Title: A Self-Controlled Study on the Treatment of Restless Legs Syndrome in Uremia With Dipyridamole
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yunfeng Xia (Other)
Responsible Party: Sponsor-Investigator, Yunfeng Xia, Chief Physician of Nephrology、Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-451-02; CYYY-SSCX202522 (Other Grant/Funding Number: The 2025 Graduate Research Innovation Project of the First Affiliated Hospital of Chongqing Medical University)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Restless Leg Syndrome Due to Uraemia
Keywords: Restless Leg Syndrome; Uraemia
MeSH Terms: conditions — Restless Legs Syndrome; Uremia | interventions — Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants will: Take dipyridamole daily (50mg each time, three times a day) for 6 months (Experimental): Participants will: Take dipyridamole daily (50mg each time, three times a day) for 6 months
  Interventions: Drug: Dipyridamole 50mg tid

INTERVENTIONS:
Drug: Dipyridamole 50mg tid — Participants will take dipyridamole daily (50mg each time, three times a day) for 6 months

SUMMARY:
The purpose of this clinical trial is to determine whether dipyridamole can treat restless legs syndrome in patients with uremia. In addition, the safety of dipyridamole will also be evaluated. The main questions this study aims to answer include: Can dipyridamole improve the symptoms of restless legs syndrome in participants? Can dipyridamole improve participants' anxiety, depression, sleep quality, and quality of life? What adverse reactions might participants experience while taking dipyridamole? This study is a self-controlled trial in which all participants receive active drug treatment. Participants will take dipyridamole daily (50 mg per dose, three times a day) for 6 months. The efficacy of dipyridamole will be evaluated by comparing relevant scale scores and laboratory indicators before and after treatment. In addition, adverse reactions during the treatment follow-up will be monitored to assess the safety of dipyridamole in this patient population.

DETAILED DESCRIPTION:
This study is a self-controlled study in which all participants received active drug treatment for 6 months. The efficacy and safety of dipyridamole were evaluated by comparing changes in relevant scale scores before and after treatment. The study screened patients receiving maintenance hemodialysis at the Hemodialysis Center of the First Affiliated Hospital of Chongqing Medical University, with a baseline score of greater than 15 on the International Restless Legs Syndrome Rating Scale (IRLS). Approximately 80 patients met the inclusion criteria of the study and were willing to sign informed consent. General clinical data and pre-study laboratory parameters were collected, including age, sex, body mass index, serum iron, ferritin, serum parathyroid hormone, hemoglobin, albumin, dialysis adequacy, IRLS, Pittsburgh Sleep Quality Index, Hamilton Depression Rating Scale, Hamilton Anxiety Rating Scale, and KDQOLTM-36. All enrolled patients were instructed to take dipyridamole tablets orally at a dose of 50 mg three times daily for 6 months. During the study, the occurrence of drug-related adverse reactions such as nausea, headache, dizziness, diarrhea, insomnia, fatigue, and bleeding was also recorded. At the end of the treatment period, general clinical data, laboratory parameters, and relevant scale assessment results were collected again.

ELIGIBILITY:
Inclusion Criteria:

(1) Maintenance hemodialysis for ≥3 months;(2) Age between 18-75 years;(3) Diagnosed with Restless Legs Syndrome (RLS) according to IRLSSG standards with a score >15;(4) Willing to cooperate with this study.

Exclusion Criteria:

(1). Patients with other cerebrovascular, muscular, and movement system diseases affecting the assessment of RLS;(2). Patients with active bleeding, such as gastrointestinal bleeding or intracerebral hemorrhage;(3). Patients who have been on dipyridamole for a long time;(4). Patients who have taken other medications that may affect RLS in the last 3 weeks, such as dopamine agonists/antagonists, tricyclic antidepressants, lithium, etc.;(5). Patients with a history of psychosis;(6). Pregnant or breastfeeding women;(7). Patients who are allergic or intolerant to dipyridamole;(8). Patients who cannot or are unwilling to cooperate with this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group rating scale | From enrollment to the end of treatment at 6 months
  The treatment effect on participants' restless legs syndrome is mainly assessed through their scores on the International Restless Legs Syndrome Study Group rating scale before and after treatment.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | From enrollment to the end of treatment at 6 months
  The changes in participants' depressive symptoms were assessed using the Hamilton Depression Rating Scale before and after they received treatment.
Hamilton Anxiety Scale | From enrollment to the end of treatment at 6 months
  The changes in participants' anxiety levels were assessed using the Hamilton Anxiety Scale before and after they received treatment.
Pittsburgh Sleep Quality Index | From enrollment to the end of treatment at 6 months
  The changes in participants' sleep quality were assessed using the Pittsburgh Sleep Quality Index before and after they received treatment.
KDQOL-36 Scale | From enrollment to the end of treatment at 6 months
  Changes in participants' quality of life were assessed using the KDQOL-36 Scale before and after they received treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided